CLINICAL TRIAL: NCT03855163
Title: Effectiveness of the Labour Inspection Authority's Regulatory Tools on Work Environment and Employee Health - Study Protocol for a Cluster Randomized Controlled Trial Among Norwegian Home-care Workers
Brief Title: Effects of Regulatory Tools on Work Environment and Employee Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Occupational Health, Norway (Other Government)
Collaborators: Norwegian Labour Inspection Authority (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201700498
Record Dates: First submitted 2019-02-15; First posted 2019-02-26 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Occupational Health; Sick Leave; Occupational Exposure
Keywords: Mental Distress; Musculoskeletal Pain; Work-related; Cluster Randomized Trial; Effect Evaluation
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: cluster-randomized controlled trial
Who Masked: Investigator
Masking Description: the study group assignment is kept hidden from the data-analysts and manuscript writers after allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inspection visits (Experimental): Regulatory tool to ensure enterprise compliance with legal requirements
  Interventions: Behavioral: Inspection visits
- Guidance workshops (Experimental): Regulatory tool applied to inform and advise enterprises on legal requirements and how to realize compliance with such requirements
  Interventions: Behavioral: Guidance workshops
- Online risk assessment tool (Experimental): Regulatory tool applied to aid enterprises in conducting written objectives concerning health, environment and safety activities
  Interventions: Behavioral: Online risk assessment tool
- Control group (No Intervention): The Labour Inspection Authority will not preform any intervention activities in enterprises assign to the control group

INTERVENTIONS:
Behavioral: Inspection visits — Normative intervention aimed at enforcing compliance with legal occupational health and safety requirements
  Arms: Inspection visits
Behavioral: Guidance workshops — Pedagogical intervention aimed to motivate managers and employee representatives to comply with legal occupational health and safety requirements
  Arms: Guidance workshops
Behavioral: Online risk assessment tool — Pedagogical intervention aimed to motivate managers and employee representatives to comply with legal occupational health and safety requirements
  Arms: Online risk assessment tool

SUMMARY:
This study evaluates the effects of the Labour Inspection Authority's regulatory tools on workplace exposures to prevent employee ill health. Norwegian municipal enterprises with employees in the home care sector have been randomized to three different experimental groups and to one control group. We hypothesize a significant lower level of work environmental exposures and health complaints, after adjusting for pre-intervention measures, in the experimental groups compared to the control group.

DETAILED DESCRIPTION:
A variety of work environmental exposures are shown to cause ill health. Compliance with occupational health and safety legislation and regulation is assumed to prevent work-related ill health. The Norwegian Labour Inspection Authority oversees that enterprises comply with the requirements of the working environment laws and regulations. The agency possesses two key regulatory tools to ensure compliance, i.e. inspections and guidance.

Inspections are used to check whether enterprises meet legal requirements. If inspectors reveal violations to legal requirements, the Labour Inspection Authority may respond with orders, coercive fines, and shutdown of operations and in worst-case report enterprises to the police.

Guidance are used to notify the enterprises of the legal requirements pertaining to work environmental standards, and to advice the employers and employee representatives concerning the most effective means of realizing compliance with the legal requirements.

Enterprises randomized to the experimental groups will receive one of three different intervention activities from the Labour Inspection Authority, i.e. targeted inspection visits, participation on a one-day workshop led by two inspectors on how to reach compliance with occupational health and safety (OHS) standards, or participation in an online risk assessment course for conducting written objectives in relation to health, environment and safety activities.

The interventions will be carried out at the organizational level (enterprise), whereas the effects of the interventions on working environment and health complaints will be measured at the individual level (employee). Two months before the Labour Inspection Authority perform their interventions, a baseline questionnaire assessing self-reported organizational, psychosocial and mechanical work factors and health complaints will be sent to all home-care workers employed in the included municipal enterprises. The effects of the different interventions on work environment and employee health will be evaluated through questionnaire measurements 6, 12 and 20 months post interventions.

ELIGIBILITY:
Inclusion Criteria:

* All employees in municipal enterprises that provide home care services with a minimum of 20 employees and a maximum of 100 employees.

Exclusion Criteria:

* Employees in municipal enterprises that have received an inspection from the Labour Inspectorate in the years 2017 and 2018.

Ages: 16 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2555 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Changes in self reported occupational exposures | Self-Reported Occupational Exposures will be assessed 2 months prior to the interventions and 12 months post interventions
  Psychosocial, organizational and mechanical factors at work will be assessed by the General Nordic Questionnaire for Psychological and Social Factors at Work (QPSNordic) and with items adapted from the following questionnaire developed by Statistics Norway: "Working environment, survey on living conditions". The wording of the questions are typically: "how often in your job do you have to … " (e.g. suppress emotions in order to appear neutral on the outside?), or "In the course of your work" ... (e.g. do you need to squat or kneel?). Level of exposure is assessed by frequency scoring on a five-point scale ranging from "1 = very seldom or never" to "5 = very often or always"
Changes in psychological distress HSCL-5 | Psychological Distress will be assessed 2 months prior to the interventions and 12 months post interventions
  Hopkins Symptom Checklist (HSCL-5), is a self-administered 5-item instrument, each item is on a four-point scale ranging from 1="not at all" to 4="extremely". Participants are asked to assess symptoms during the past 2 weeks prior to answering the questionnaire. The average item score is calculated by dividing the total score of the number of items answered (ranging between 1.00 and 4.00).
Changes in musculoskeletal pain | Musculoskeletal Pain will be assessed 2 months prior to the interventions and 12 months post interventions
  Self-reported intensity of pain in five anatomic sites; neck, shoulder, back, arm, and leg. Each question is phrased: "Have you been troubled by… (e.g. neck pain) the last 4 weeks? Response alternatives are: 1) "not troubled", 2) "a little troubled", 3) "rather intensely troubled" and 4)" very intensely troubled"
Changes in physician-certified absence from work, number of events (17 days or more) per 100 employee-years | The absence rate will be assessed during the one year prior to the interventions and during the one year after the interventions
  Data from the Norwegian Labour and Welfare Administration's sickness benefit register. This register provides complete registrations of all sickness absence episodes-including the length and medical diagnosis-which are compensated by the national insurance sickness benefit. As a general rule, everybody working or living in Norway is covered by the Norwegian national social insurance.

CONTACTS AND LOCATIONS:
Overall Officials: Håkon A Johannessen, PhD, Principal Investigator — National Institute of Occupational Health
Locations (130):
- Norway (130):
  - Hjemmetjenesten i Tysvær kommune, Tysvær, Aksdal
  - Hjemmetjenesten i Averøy kommune, Vebenstad, Averøy
  - Hjemmetjenesten i Evenes kommune, Evenes, Bogen
  - Hjemmetjenesten i Dønna kommune, Dønnes, Dønna
  - Hjemmetjenesten i Åsnes kommune, Åsnes, Flisa
  - Hjemmetjenesten i Luster kommune, Luster, Gaupne
  - Hjemmetjenesten i Nannestad kommune, Teigebyen, Nannestad
  - Hjemmetjenesten i Storfjord kommune, Storfjord, Oteren
  - Hjemmetjenesten i Åmot kommune, Åmot, Rena
  - Hjemmetjenesten i Rendalen kommune, Redalen, Rendalen
  - Hjemmetjenesten i Råde kommune, Moss, Råde
  - Hjemmetjenesten i Gloppen kommune, Vereide, Sandane
  - Hjemmetjenesten i Skjåk kommune, Skår, Skjåk
  - Hjemmetjenesten i Sund kommune, Sund, Skogsvåg
  - Hjemmetjenesten i Smøla kommune, Smørås, Smøla
  - Hjemmetjenesten i Stord kommune, Leirvik, Stord
  - Hjemmetjenesten i Trøgstad kommune, Mysen, Trøgstad
  - Hjemmetjenesten i Giske kommune, Ålesund, Valderøya
  - Hjemmetjenesten i Vang kommune, Vang, Valdres
  - Hjemmetjenesten i Vega kommune, Nordland, Vega
  - Hjemmetjenesten i Lindesnes kommune, Linnes, Vest-Agder
  - Hjemmetjenesten i Andøy kommune, Andenes
  - Hjemmetjenesten i Askvoll kommune, Askvoll
  - Hjemmetjenesten i Aure kommune, Aure
  - Hjemmetjenesten i Aurland kommune, Aurland
  - Hjemmetjenesten i Ål kommune, Ål
  - Hjemmetjenesten i Åmli kommune, Åmli
  - Hjemmetjenesten i Årdal kommune, Årdalstangen
  - Hjemmetjenesten i Ballangen kommune, Ballangen
  - Hjemmetjenesten i Aurskog Høland kommune, Bjørkelangen
  - Hjemmetjenesten i Kvæfjord kommune, Borkenes
  - Hjemmetjenesten i Haram kommune, Brattvåg
  - Hjemmetjenesten i Hasvik kommune, Breivikbotn
  - Hjemmetjenesten i Time kommune, Bryne
  - Hjemmetjenesten i Kvænangen kommune, Burfjord
  - Hjemmetjenesten i Bø, Bø
  - Hjemmetjenesten i Nordre Land kommune, Dokka
  - Hjemmetjenesten i Drammen kommune, Drammen
  - Hjemmetjenesten i Drangedal kommune, Drangedal
  - Hjemmetjenesten i Frogn kommune, Drøbak
  - Hjemmetjenesten i Eide kommune, Eide
  - Hjemmetjenesten i Gulen kommune, Eivindvik
  - Hjemmetjenesten i Elverum kommune, Elverum
  - Hjemmetjenesten i Skånland kommune, Evenskjer
  - Hjemmetjenesten i Evje og Hornnes kommune, Evje
  - Hjemmetjenesten i Nord-Aurdal kommune, Fagernes
  - Hjemmetjenesten i Fauske kommune, Fauske
  - Hjemmetjenesten i Fedje kommune, Fedje
  - Hjemmetjenesten i Flekkefjord kommune, Flekkefjord
  - Hjemmetjenesten i Herøy kommune, Fosnavåg
  - Hjemmetjenesten i Fyresdal kommune, Fyresdal
  - Hjemmetjenesten i Gjerstad kommune, Gjerstad
  - Hjemmetjenesten i Gol kommune, Gol
  - Hjemmetjenesten i Hareid kommune, Hareid
  - Hjemmetjenesten i Øvre Eiker kommune, Hokksund
  - Hjemmetjenesten i Søndre Land kommune, Hov
  - Hjemmetjenesten i Ringerike kommune, Hønefoss
  - Hjemmetjenesten i Iveland kommune, Iveland
  - Hjemmetjenesten i Ullensaker kommune, Jessheim
  - Hjemmetjenesten i Jevnaker kommune, Jevnaker
  - Hjemmetjenesten i Strand kommune, Jørpeland
  - Hjemmetjenesten i Grue kommune, Kirkenær
  - Hjemmetjenesten i Klepp kommune, Kleppe
  - Hjemmetjenesten i Hemnes kommune, Korgen
  - Hjemmetjenesten i Kragerø kommune, Kragerø
  - Hjemmetjenesten i Kvinesdal kommune, Kvinesdal
  - Hjemmetjenesten i Bamble kommune, Langesund
  - Hjemmetjenesten i Sande kommune Møre og Romsdal, Larsnes
  - Hjemmetjenesten i Leikanger kommune, Leikanger
  - Hjemmetjenesten i Steigen kommune, Leinesfjorden
  - Hjemmetjenesten i Leirfjord kommune, Leirfjord
  - Hjemmetjenesten i Vestvågøy kommune, Leknes
  - Hjemmetjenesten i Lesja kommune, Lesja
  - Hjemmetjenesten i Lillesand, Lillesand
  - Hjemmetjenesten i Osterøy kommune, Lonevåg
  - Hjemmetjenesten i Lærdal kommune, Lærdal
  - Hjemmetjenesten i Løten kommune, Løten
  - Hjemmetjenesten i Midsund kommune, Midsund
  - Hjemmetjenesten i Rana kommune, Mo i Rana
  - Hjemmetjenesten i Målselv kommune, Moen
  - Hjemmetjenesten i Vefsen kommune, Mosjøen
  - Hjemmetjenesten i Eidsberg kommune, Mysen
  - Hjemmetjenesten i Nes kommune Buskerud, Nesbyen
  - Hjemmetjenesten i Songdalen kommune, Nodeland
  - Hjemmetjenesten i Kvam kommune, Norheimsund
  - Hjemmetjenesten i Notodden kommune, Notodden
  - Hjemmetjenesten i Odda kommune, Odda
  - Hjemmetjenesten i Sel kommune, Otta
  - Hjemmetjenesten i Sigdal kommune, Prestfoss
  - Hjemmetjenesten i Rakkestad kommune, Rakkestad
  - Randaberg kommune, Randaberg
  - Hjemmetjenesten i Re kommune, Re
  - Hjemmetjenesten i Risør kommune, Risør
  - Hjemmetjenesten i Tinn kommune, Rjukan
  - Hjemmetjenesten i Kvinnherad kommune, Rosendal
  - Hjemmetjenesten i Lunner kommune, Røa
  - Hjemmetjenesten i Nore og Uvdal kommune, Rødberg
  - Hjemmetjenesten i Hole kommune, Røyse
  - Hjemmetjenesten i Nord-Odal kommune, Sagstua
  - Hjemmetjenesten i Suldal kommune, Sand
  - Hjemmetjenesten i Sauda kommune, Sauda
  - Hjemmetjenesten i Hjartdal kommune, Sauland
  - Hjemmetjenesten i Selje kommune, Selje
  - Hjemmetjenesten i Seljord kommune, Seljord
  - Hjemmetjenesten i Sør-Odal kommune, Skarnes
  - Hjemmetjenesten i Hvaler kommune, Skjærhalden
  - Hjemmetjenesten i Sola kommune, Sola
  - Hjemmetjenesten i Spydeberg kommune, Spydeberg
  - Hjemmetjenesten i Stordal kommune, Stordal
  - Hjemmetjenesten i Nordreisa kommune, Storslett
  - Hjemmetjenesten i Sørfold kommune, Straumen
  - Hjemmetjenesten i Bø kommune Nordland, Straumsjøen
  - Hjemmetjenesten i Sunndal kommune, Sunndalsøra
  - Hjemmetjenesten i Sveio kommune, Sveio
  - Hjemmetjenesten i Vågan kommune, Svolvær
  - Hjemmetjenesten i Sykkylven kommune, Sykkylven
  - Hjemmetjenesten i Sørreisa kommune, Sørreisa
  - Hjemmetjenesten i Tvedestrand kommune, Tvedestrand
  - Hjemmetjenesten i Tynset kommune, Tynset
  - Hjemmetjenesten i Samnanger kommune, Tysse
  - Hjemmetjenesten i Tysnes kommune, Uggdal
  - Hjemmetjenesten i Vennesla kommune, Vennesla
  - Hjemmetjenesten i Vinje kommune, Vinje
  - Hjemmetjenesten i Nord-Fron kommune, Vinstra
  - Hjemmetjenesten i Volda kommune, Volda
  - Hjemmetjenesten i Vindafjord kommune, Ølen
  - Hjemmetjenesten i Marker kommune, Ørje
  - Hjemmetjenesten i Meløy kommune, Ørnes
  - Hjemmetjenesten i Gausdal kommune, Østre Gausdal
  - Hjemmetjenesten i Øyer kommune, Øyer

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available 3 years after study completion
Access Criteria: Data access request will be reviewed by NSD - Norwegian Centre for Research Data
URL: https://nsd.no/nsd/english/index.html

REFERENCES:
- [Background] M. Dallner, A.-L. Elo, F. Gamberale, V. Hottinen, S. Knardahl, K. Lindström, A. Skogstad, E. Ørhede. Validation of the General Nordic Questionnaire (QPSNordic) for psychological and social factors at work. Nordic Council of Ministers, Copenhagen (2000)
- [Background] Christensen JO, Nielsen MB, Finne LB, Knardahl S. Comprehensive profiles of psychological and social work factors as predictors of site-specific and multi-site pain. Scand J Work Environ Health. 2018 May 1;44(3):291-302. doi: 10.5271/sjweh.3706. Epub 2018 Jan 11. PMID 29325179
- [Background] Andersen JH, Malmros P, Ebbehoej NE, Flachs EM, Bengtsen E, Bonde JP. Systematic literature review on the effects of occupational safety and health (OSH) interventions at the workplace. Scand J Work Environ Health. 2019 Mar 1;45(2):103-113. doi: 10.5271/sjweh.3775. Epub 2018 Oct 29. PMID 30370910
- [Background] Mischke C, Verbeek JH, Job J, Morata TC, Alvesalo-Kuusi A, Neuvonen K, Clarke S, Pedlow RI. Occupational safety and health enforcement tools for preventing occupational diseases and injuries. Cochrane Database Syst Rev. 2013 Aug 30;2013(8):CD010183. doi: 10.1002/14651858.CD010183.pub2. PMID 23996220
- [Background] Strand BH, Dalgard OS, Tambs K, Rognerud M. Measuring the mental health status of the Norwegian population: a comparison of the instruments SCL-25, SCL-10, SCL-5 and MHI-5 (SF-36). Nord J Psychiatry. 2003;57(2):113-8. doi: 10.1080/08039480310000932. PMID 12745773
- [Background] Stromholm T, Pape K, Ose SO, Krokstad S, Bjorngaard JH. Psychosocial working conditions and sickness absence in a general population: a cohort study of 21,834 workers in Norway (The HUNT Study). J Occup Environ Med. 2015 Apr;57(4):386-92. doi: 10.1097/JOM.0000000000000362. PMID 25851186
- [Derived] Knutsen RH, Nielsen MB, Lunde LK, Fostervold KI, Johannessen HA. Sick leave due to musculoskeletal disorders: A prospective cohort study. Int J Nurs Stud Adv. 2025 Jul 6;9:100376. doi: 10.1016/j.ijnsa.2025.100376. eCollection 2025 Dec. PMID 40851813
- [Derived] Johannessen HA, Knardahl S, Emberland JS, Skare O, Finnanger Garshol B. Do regulatory tools instigate measures to prevent work-related psychosocial and ergonomic risk factors? A process evaluation of a Labour inspection authority trial in the Norwegian home-care services. BMC Res Notes. 2022 Nov 18;15(1):349. doi: 10.1186/s13104-022-06244-4. PMID 36401320
- [Derived] Finnanger Garshol B, Knardahl S, Emberland JS, Skare O, Johannessen HA. Effects of the Labour Inspectorate Authority's regulatory tools on psychosocial and biomechanical work factors in Norwegian home care services: a cluster randomised controlled trial. Occup Environ Med. 2022 Dec;79(12):807-815. doi: 10.1136/oemed-2022-108470. Epub 2022 Sep 27. PMID 36167785
- [Derived] Indregard AR, Knardahl S, Emberland JS, Skare O, Johannessen HA. Effectiveness of the Labour Inspection Authority's regulatory tools for work environment and employee health: study protocol for a cluster-randomised controlled trial among Norwegian home-care workers. BMJ Open. 2019 Nov 26;9(11):e031226. doi: 10.1136/bmjopen-2019-031226. PMID 31772092
- See also: Statistics Norway, Working environment, survey on living conditions — https://www.ssb.no/en/arbeid-og-lonn/statistikker/arbmiljo